CLINICAL TRIAL: NCT02918110
Title: Vaginal Misodel® in Comparison With Orally Administrated Misoprostol (Cytotec®) at Induction of Labour
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Karlstad Central Hospital (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1cyt
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Induced Deliveries
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytotec (Experimental): orally administrated solution of misoprostol (Cytotec®)
  Interventions: Drug: Misoprostol
- Misodel (Experimental): vaginal slow release misoprostol (Misodel®)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Women needed to be induced will get orally administrated solution of misoprostol (Cytotec®) or vaginal slow release misoprostol (Misodel®)
  Other Names: Cytotec

SUMMARY:
The study will compare orally administrated solution of Misoprostol (Cytotec®) with vaginal slow release (7ug/h) Misoprostol (Misodel®) regarding efficacy and safety during labour.

DETAILED DESCRIPTION:
To compare orally administrated solution of misoprostol (Cytotec®) with vaginal slow release misoprostol (Misodel®) regarding efficacy and safety during labour Design: Randomised controlled trial (RCT)

Settings:

Obstetric departments of Sodersjukhuset, Stockholm Obstetric departments of Women's clinic, Karlstad.

ELIGIBILITY:
Inclusion Criteria:

Primipara BS ≤ 4p Gestational week >37

Exclusion Criteria:

Multipara Multiples Gestational week <37 BS >4 IUFD Previous uterine surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Cesarean section rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Per Tornvall, Prof, Study Director — Karolinska Institutet
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strandberg M, Wallstrom T, Wiberg-Itzel E. Women's expectations and experiences of labor induction - a questionnaire-based analysis of a randomized controlled trial. BMC Pregnancy Childbirth. 2021 May 4;21(1):355. doi: 10.1186/s12884-021-03786-6. PMID 33947349